CLINICAL TRIAL: NCT01086800
Title: Phase II Trial of Sleep Apnea Treatment to Reduce Cardiovascular Morbidity
Brief Title: Heart Biomarker Evaluation in Apnea Treatment
Acronym: HeartBEAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Case Western Reserve University (Other); Partners HealthCare (Other); Johns Hopkins University (Other); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Redline, Senior Physician, Division of Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1RC2HL101417-01 (NIH)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Cardiovascular Disease; Obstructive Sleep Apnea; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Sleep Apnea, Obstructive; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HLSE plus PAP (Other)
  Interventions: Other: Healthy Lifestyles and Sleep Education plus PAP
- HLSE plus Oxygen (Other)
  Interventions: Other: Healthy Lifestyles and Sleep Education plus Supplemental Oxygen
- Healthy Lifestyles and Sleep Education (Other)
  Interventions: Other: Healthy Lifestyles and Sleep Education

INTERVENTIONS:
Other: Healthy Lifestyles and Sleep Education plus PAP — Participants randomized to this arm will be educated on PAP and then use PAP for 3 months. They will also receive optimized medical preventive therapy according to current American Heart Association guidelines for prevention of CVD and sleep guidelines.
  Arms: HLSE plus PAP
Other: Healthy Lifestyles and Sleep Education plus Supplemental Oxygen — Participants randomized to this arm will be educated on nocturnal supplemental oxygen and then use oxygen for 3 months. They also will receive optimized medical preventive therapy according to current American Heart Association guidelines for prevention of CVD and sleep guidelines.
  Arms: HLSE plus Oxygen
Other: Healthy Lifestyles and Sleep Education — Participants randomized to this arm will receive optimized medical preventive therapy according to current American Heart Association guidelines for prevention of CVD and sleep guidelines.
  Arms: Healthy Lifestyles and Sleep Education

SUMMARY:
This study examines the role of sleep apnea treatment in improving cardiovascular biomarkers.

DETAILED DESCRIPTION:
This is a Phase II randomized controlled trial that will evaluate the effects of supplemental nocturnal oxygen or Positive Airway Pressure (PAP) therapy, compared to optimal medical preventive therapy for Cardiovascular Disease (CVD) risk, on biomarkers of CVD risk in Obstructive Sleep Apnea (OSA) patients at high risk for CVD events. The study will focus on patients with moderate to severe OSA but only mild OSA symptoms.

Eligible participants have a history or symptoms of heart disease AND have symptoms of sleep apnea or snoring. Participants will be contributing to medical knowledge about different options that can be used to improve heart disease in people with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* established Coronary Artery Disease or established cardiovascular disease risk factors
* home sleep test that showed moderately severe sleep apnea

Exclusion Criteria:

* poorly controlled health
* currently using supplemental oxygen or PAP for OSA

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To compare the effects of nocturnal supplemental oxygen and PAP versus optimized medical management on biomarkers of cardiovascular risk, including: | 3 months
  * 24 hour blood pressure (BP) profile
  * Markers of systemic inflammation
  * Markers of oxidative stress
  * Prothrombotic markers
  * Sympathetic nervous system activity
  * Cardiac rhythm, impulse generation and ischemia
  * Dyslipidemia
  * Glucose regulation
  * Myocardial stress

SECONDARY OUTCOMES:
Compare the effects of nocturnal supplemental oxygen and PAP versus standard care on patient-reported outcomes, including: | 3 months
  * vitality
  * self reported sleepiness
Compare nocturnal supplemental oxygen and PAP on measures of: | 3 months
  * efficacy (AHI, hypoxemia)
  * adherence
  * side effects

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Partners HealthCare, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Hilmisson H, Thomas RJ, Magnusdottir S. Cardiopulmonary coupling-calculated sleep stability and nocturnal heart rate kinetics as a potential indicator for cardiovascular health: a relationship with blood pressure dipping. Front Sleep. 2024 Aug 1;3:1230958. doi: 10.3389/frsle.2024.1230958. eCollection 2024. PMID 41424523
- [Derived] Ni YN, Lei F, Tang X, Liang Z, Thomas RJ. The association between the effective apnea-hypopnea index and blood pressure reduction efficacy following CPAP/oxygen treatment. Sleep Med. 2024 May;117:46-52. doi: 10.1016/j.sleep.2024.02.046. Epub 2024 Mar 13. PMID 38507976
- [Derived] Schmickl CN, Orr JE, Sands SA, Alex RM, Azarbarzin A, McGinnis L, White S, Mazzotti DR, Nokes B, Owens RL, Gottlieb DJ, Malhotra A. Loop Gain as a Predictor of Blood Pressure Response in Patients Treated for Obstructive Sleep Apnea: Secondary Analysis of a Clinical Trial. Ann Am Thorac Soc. 2024 Feb;21(2):296-307. doi: 10.1513/AnnalsATS.202305-437OC. PMID 37938917
- [Derived] Magnusdottir S, Thomas RJ, Hilmisson H. Can improvements in sleep quality positively affect serum adiponectin-levels in patients with obstructive sleep apnea? Sleep Med. 2021 Aug;84:324-333. doi: 10.1016/j.sleep.2021.05.032. Epub 2021 May 29. PMID 34225174
- [Derived] Magnusdottir S, Hilmisson H, Thomas RJ. Cardiopulmonary coupling-derived sleep quality is associated with improvements in blood pressure in patients with obstructive sleep apnea at high-cardiovascular risk. J Hypertens. 2020 Nov;38(11):2287-2294. doi: 10.1097/HJH.0000000000002553. PMID 32649638
- [Derived] Gottlieb DJ, Punjabi NM, Mehra R, Patel SR, Quan SF, Babineau DC, Tracy RP, Rueschman M, Blumenthal RS, Lewis EF, Bhatt DL, Redline S. CPAP versus oxygen in obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2276-85. doi: 10.1056/NEJMoa1306766. PMID 24918372